CLINICAL TRIAL: NCT02515149
Title: Randomized Controlled Trial to Assess Accuracy, Feasibility, Acceptability, Cost Effectiveness and Impact of Point of Care CD4 Testing on HIV Diagnosis, Linkage to Care and Time to Antiretroviral Therapy Initiation Among HIV Infected Patients in Rural Western Kenya
Brief Title: Impact on Linkage to HIV Care With Point of Care CD4 Testing and Home-based HIV Testing in Kenya
Acronym: CD4-POC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Kenya Medical Research Institute (Other); United States President's Emergency Plan for AIDS Relief (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CDC - NCHHSTP - 6382
Record Dates: First submitted 2015-08-03; First posted 2015-08-04 (Estimated); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: HIV
Keywords: linkage to care; point of care diagnostics; point of care CD4; HIV care cascade; Kenya

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care (No Intervention): Referral laboratory based CD4 measurement after home-based HIV testing
- Point of care (Experimental): POC CD4 testing after home-based HIV testing
  Interventions: Device: Point of care CD4 device (Alere PIMA)

INTERVENTIONS:
Device: Point of care CD4 device (Alere PIMA) — for persons testing + with home-based HIV testing using Kenya's two rapid test algorithm, intervention arm participants received point of care CD4 testing followed by counseling on results which included their treatment eligibility
  Other Names: Alere Pima
  Arms: Point of care

SUMMARY:
Randomised Controlled Trial to Assess Accuracy, Feasibility, Acceptability, Cost Effectiveness and Impact of Point of Care CD4 Testing on HIV Diagnosis, Linkage to Care and Time to Antiretroviral Therapy Initiation among HIV Infected Patients in Rural Western Kenya.

ELIGIBILITY:
Inclusion Criteria: adults living in the study catchment area (Gem Village, Nyanza province Western Kenya) served by one of 23 HIV clinics and 3 referral labs

* Not having received HIV care in prior 6 months if known HIV+

Exclusion Criteria:

* current HIV care or HIV care within last six months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 770 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Linkage to HIV care | Within six months from date of study enrollment
  As ascertained from clinic charts
ART initiation | Within six months from date of study enrollment
  As ascertained from clinic charts

CONTACTS AND LOCATIONS:
Locations (1):
- CDC - KEMRI Field Research Station, Kisumu, Nyanza, Kenya

REFERENCES:
- [Derived] Desai MA, Okal DO, Rose CE, Ndivo R, Oyaro B, Otieno FO, Williams T, Chen RT, Zeh C, Samandari T. Effect of point-of-care CD4 cell count results on linkage to care and antiretroviral initiation during a home-based HIV testing campaign: a non-blinded, cluster-randomised trial. Lancet HIV. 2017 Sep;4(9):e393-e401. doi: 10.1016/S2352-3018(17)30091-7. Epub 2017 May 31. PMID 28579225